CLINICAL TRIAL: NCT04624893
Title: A Multicenter, Retrospective Observational Study to Evaluate the Effectiveness and Safety of Polatuzumab Vedotin in the Treatment of Patients With Transplantation Ineligible Relapsed/Refractory Diffuse Large B-Cell Lymphoma
Brief Title: A Multicenter, Retrospective Observational Study to Evaluate the Effectiveness and Safety of Polatuzumab Vedotin
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jiangsu Cancer Institute & Hospital (Other)
Responsible Party: Principal Investigator, Jianqiu Wu, Director of lymphoma department, Jiangsu Cancer Institute & Hospital
Other Study IDs: PolaCUP
Record Dates: First submitted 2020-11-05; First posted 2020-11-12 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Diffuse Large B-Cell Lymphoma (DLBCL)
Keywords: Diffuse Large B-Cell Lymphoma (DLBCL); Polatuzumab Vedotin
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — polatuzumab vedotin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pola BR/R: Patients with R/R DLBCL who are enrolled in the Pola CUP program in China, and treated with Pola-BR or Pola-R regimens.
  Interventions: Drug: Polatuzumab Vedotin-Piiq

INTERVENTIONS:
Drug: Polatuzumab Vedotin-Piiq — Patients will receive a total of six cycles of Pola in combination with rituximab and bendamustine or in combination with only rituximab. A cycle is typically 21 days for DLBCL.
  Other Names: Polatuzumab Vedotin

SUMMARY:
To assess the clinical outcomes following treatment with Pola in combination with Bendamustine, Rituximab (BR) or Rituximab (R) in patients with R/R DLBCL who are not eligible for transplantation in the real-world setting.

DETAILED DESCRIPTION:
This study is a multi-center retrospective observational study. It aims to evaluate the effectiveness and safety of polatuzumab vedotin treatment in patients with hematopoietic stem cell transplantation ineligible relapsed/refractory diffuse large B-cell lymphoma (R/R DLBCL), who met the criteria to access Pola through the compassionate use program (CUP). Based on the medical records of patients in the four participating hospitals, the study database will be established by using the unified case report form (CRF) to search extract information the data of target population from the hospital database, that is, the variables without personal identification information.

ELIGIBILITY:
Inclusion Criteria:

Hospitalized patients Patients who enrolled in the Pola CUP program and met the following criteria:

* Histologically confirmed DLBCL, patients have exhausted all therapeutic options for DLBCL and have been treated with at least two prior lines of therapy including R-CHOP (or similar regimen for 1L DLBCL)
* Not considered to be eligible for Bone Marrow Transplantation (BMT) (both allogenic or autologous)
* Have documented recent progression following or during last treatment, or became intolerant to the last treatment
* Does not have ≥ Grade 2 peripheral neuropathy(PN) prior to receiving Pola
* Patients treated with Pola-BR or Pola-R regimens

Exclusion Criteria:

* Patients participating in other clinical studies of Pola.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients enrolled in the Pola CUP program in China
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2019-12-12 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Investigator-assessed best overall response (BOR) | From the start of the treatment until the date of first documented progression or the completion of the treatment(up to six cycles, each cycle is 21 days)
  Best overall response (BOR) assessed by the investigator, is based on either PET-CT or CT, and defined as the percentage of patients with CR or PR.

SECONDARY OUTCOMES:
Objective response rate (ORR) | At end of the treatment(up to six cycles, each cycle is 21 days)
  Objective response rate (ORR) assessed by the investigator at the end of treatment (EOT), is defined as the percentage of patients with CR or PR at the end of treatment.
Duration of response (DOR) | From initial CR or PR to disease progression, relapse, or death from any cause, whichever occurred first, assessed up to 25 months
  DOR is defined as the time from initial complete response (CR) or partial response (PR) to disease progression, relapse, or death from any cause, whichever occurred first.
Complete response (CR) | At end of the treatment(up to six cycles, each cycle is 21 days)
  CR rate is defined as the percentage of patients with CR.
Progression free survival (PFS) | From the start of treatment until disease progression, relapse, or death from any cause, whichever occurred first,assessed up to 30 months
  PFS is defined as the time from the start of treatment until disease progression, relapse, or death from any cause, whichever occurred first.

CONTACTS AND LOCATIONS:
Overall Officials: Jifeng Feng, Ph.D, Principal Investigator — Jiangsu Cancer Institute & Hospital
Locations (1):
- Jiangsu Cancer Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided